CLINICAL TRIAL: NCT02607527
Title: Annular Reshaping of the Mitral Valve for Patients With Mitral Regurgitation Using the Millipede IRIS System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-002, CP-003
Record Dates: First submitted 2015-10-28; First posted 2015-11-18 (Estimated); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device Implantation (Other): Transcatheter IRIS placement
  Interventions: Device: Mitral Valve IRIS Ring

INTERVENTIONS:
Device: Mitral Valve IRIS Ring — Transcatheter implantation of the IRIS

SUMMARY:
Multi center evaluation of the Millipede IRIS for treatment of clinically significant mitral regurgitation in subjects determined appropriate for mitral valve surgery.

DETAILED DESCRIPTION:
Multi center evaluation of the Millipede IRIS for treatment of clinically significant mitral regurgitation in subjects determined appropriate for mitral valve surgery.

This trial is designed in accordance with the 2014 ACC/AHA guidelines for valvular heart disease, and the consensus statement of MVARC 2015.

Subjects will undergo transcatheter implantation of the Millipede IRIS implant.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic severe MR (effective regurgitant orifice (ERO) ≥0.2 cm2 for Secondary MR, ERO ≥0.4 cm2 for Primary MR)
* The New York Heart Association Functional Class II, III or ambulatory IV.
* Left Ventricular Ejection Fraction (LVEF) is ≥20% and ≤50%
* Creatine Kinase-MB (CK-MB) obtained within prior 14 days < local laboratory -Upper Limit of Normal (ULN).
* Left Ventricular End Systolic Dimension (LVESD) is ≤ 65 mm assessed by TTE obtained within 90 days Exclusion Criteria: -Untreated clinically significant coronary artery disease requiring revascularization.

Presence of any of the following:

* Estimated pulmonary artery systolic pressure (PASP) > 70 mmHg assessed by site based on echocardiography or right heart catheterization
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
* Hemodynamic instability requiring inotropic support or mechanical heart assistance.
* Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
* Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction.
* Coronary artery bypass grafting (CABG) within 30 days prior to subject's consent.
* Percutaneous coronary intervention within 30 days prior to subject's consent.
* Tricuspid valve disease requiring surgery.
* Aortic valve disease requiring surgery or TAVI.
* Carotid surgery within 30 days prior to subject registration.
* Implant of any Cardiac Resynchronization Therapy (CRT) or Cardiac -Resynchronization Therapy with cardioverter-defibrillator (CRT-D) within the last 30 days prior to subject registration.
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months.
* Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure.
* Status 1 heart transplant or prior orthotopic heart transplantation.
* Chronic Kidney Disease.
* Chronic Steroid Therapy.
* Cerebrovascular accident within 30 days prior to subject's consent.
* Severe symptomatic carotid stenosis (> 70% by ultrasound).Life expectancy < 12 months due to non-cardiac conditions.
* Active infections requiring current antibiotic therapy.
* Pregnant or planning pregnancy within next 12 months.
* Currently participating in an investigational drug or another device study.
* Severe organic lesions with mitral chords retraction, severely fibrotic and immobile leaflets, severely deformed subvalvular apparatus.
* endocarditis or active endocarditis in the last 3 months.
* Heavily calcified annulus or leaflets, mitral valve stenosis.
* Congenital malformation with limited valvular tissue
* Patient requires mitral valve replacement
* Previously implanted prosthetic mitral valve or annuloplasty ring/band.
* Evidence of LV or LA thrombus, vegetation or mass
* Left Ventricular Ejection Fraction <20%
* Left Ventricular End Diastolic Diameter >65 mm
* Severe tricuspid regurgitation or severe RV dysfunction
* Condition that prevents transatrial access or transfemoral access
* Anatomical ineligibility to the investigational device
* Known hypersensitivity or contraindication to procedural or post procedural medication (e.g., contrast solution, anticoagulation therapy) or hypersensitivity to nickel or titanium.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Acute Safety defined as incidence of adverse events | Procedure through 30 days post procedure
  30 days defined as ability to implant, anchor and actuate without incidence of adverse events

SECONDARY OUTCOMES:
Efficacy assessed by reduction in mitral regurgitation without significant mitral stenosis as measured by echo | Procedural through 48 hrs post procedure
  Reduction in mitral regurgitation to optimal or acceptable levels without significant mitral stenosis post procedure (defined as discharge or 48 hrs whichever comes first) and EROA <1.5 cm2 with transmitral gradient <5mm Hg as compared to screening echo

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Dante Pazzanese de Cardiologia
Locations (2):
- Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided